CLINICAL TRIAL: NCT04383171
Title: A Prospective Observational Cohort Study - Does Early Limb Ergometry Affect Oxygen Delivery and Uptake in Intubated Critically Ill Patients?
Brief Title: Looking at the Physiological Response of Ergometry in Critical Care Patients
Status: Completed | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: southamptonNHSTrust
Record Dates: First submitted 2019-12-11; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2019-12

CONDITIONS: Critical Ill Patients
Keywords: Early rehabilitation; Physiological response; Critical care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: Motomed cycle ergometer (MOTOmed letto2 - Reck, Reckstr 1-5, Betzenweiler 88422, Germany).

SUMMARY:
Exploring the physiological and metabolic demands of passive ergometry in the critical ill patient.

DETAILED DESCRIPTION:
This study explores the physiological and metabolic demands of passive ergometry as a step in active rehabilitation and compares two methods of monitoring these changes in critically ill patients.

ELIGIBILITY:
Inclusion Criteria

* already on the Early Mobility Programme (EMP)
* cardiovascularly stable (stable vasopressor dose for two hours)
* stable heart rate (<140 bpm) and heart rhythm
* presence of a jugular central venous pressure (CVP) line and arterial line.

Exclusion Criteria

* prior rapidly deteriorating neuromuscular disease
* upper limb problem precluding cycle ergometry
* pyrexia (temp >38 °C)
* raised intracranial pressure
* poor prognostic outcomes
* lack of agreement from clinician
* Next of kin/Legal representative (NOK/LR) not understanding English.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All adult patients admitted to the Intensive Care Unit with a medical diagnosis and requiring intubation and ventilation for at least 48 hours and on the Early Mobility Programme (EMP) within 72 hours of admission.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2015-03-17 (Actual); Primary Completion 2017-06-07 (Actual); Study Completion 2017-06-07 (Actual)

PRIMARY OUTCOMES:
Physiological demands of early passive ergometry use in the critically ill patient. | Minute by minute measurements were taken over the 60 minute data collection period.
  Haemodynamic measurements collected were arterial systolic and diastolic blood pressure (SBP/DBP mmHg).
Physiological demands of early passive ergometry use in the critically ill patient. | Minute by minute measurements were taken over the 60 minute data collection period.
  Haemodynamic measurements collected were heart rate (HR beats/min).
Physiological demands of early passive ergometry use in the critically ill patient. | Minute by minute measurements were taken over the 60 minute data collection period.
  Haemodynamic measurements collected were cardiac output (CO L/min).
Physiological demandsof early passive ergometry use in the critically ill patient. | Minute by minute measurements were taken over the 60 minute data collection period.
  Respiratory measurements collected were stroke volume (SV m/L).
Physiological demands of early passive ergometry use in the critically ill patient. | Minute by minute measurements were taken over the 60 minute data collection period.
  Respiratory measurements collected were respiratory rate (RR breaths/min).
Physiological demands of early passive ergometry use in the critically ill patient. | Minute by minute measurements were taken over the 60 minute data collection period.
  Respiratory measurements collected were minute volume (MV L/min) and tidal volume (VT L/min).
Physiological demands of early passive ergometry use in the critically ill patient. | Minute by minute measurements were taken over the 60 minute data collection period.
  Metabolic measurements collected were oxygen delivery (DO2 m/L) and oxygen uptake (VO2 m/L).
Physiological demands of early passive ergometry use in the critically ill patient. | Minute by minute measurements were taken over the 60 minute data collection period.
  Metabolic measurements collected were central venous oxygen saturation (ScvO2 %).
Physiological demands of early passive ergometry use in the critically ill patient. | Minute by minute measurements were taken over the 60 minute data collection period.
  Metabolic measurements collected were CO2 production (VCO2 mL/min).
Physiological demands of early passive ergometry use in the critically ill patient. | These were taken every 10 minutes over the 60 minute data collection period.
  Paired venous and arterial blood gas samples were collected.

SECONDARY OUTCOMES:
Comparing two methods of measuring oxygen uptake (VO2 mL/min) and oxygen delivery (DO2 mL/min) during one passive ergometry session in the critically ill patient. | Minute by minute haemodynamic and metabolic measurements were taken over the 60 minute data collection period. Paired venous and arterial blood gas samples were taken every 10 minutes over the 60 minute data collection period.
  Oxygen uptake (VO2) was calculated by two methods.
  1. Method one calculated VO2 with the value of CO from the LiDCO™ using the modified technique of the Fick equation using paired central mixed venous and arterial blood gas samples: VO2 mL/min = CO x (CaO2 - CvO2) x10.
  2. Method two calculated VO2 by the E-COVX metabolic module via the ventilator from the value of fraction of inspired O2 (FiO2), expiratory minute volume (MV), expired concentrations of O2 (FeO2) and CO2 (FeCO2) using the equation: VO2 ml/min= MV (FiO2 -FeO2 - FiO2 (FeCO2))/1-FiO2.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wilkinson OM, Bates A, Cusack R. An observational feasibility study - does early limb ergometry affect oxygen delivery and uptake in intubated critically ill patients - a comparison of two assessment methods. BMC Anesthesiol. 2021 Jan 25;21(1):27. doi: 10.1186/s12871-020-01227-z. PMID 33494702